CLINICAL TRIAL: NCT07279376
Title: Harnessing Data Science to Improve HIV Care Continuum Outcomes: A Hybrid Type 2 Trial Evaluating a Machine-Learning Algorithm-Based Implementation Strategy
Brief Title: Evaluating an Algorithm-Based Implementation Strategy to Improve HIV Care Outcomes
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter College of City University of New York (Other)
Responsible Party: Principal Investigator, Sarit Golub, Distinguished Professor, Hunter College of City University of New York
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: R01MH136903 (NIH)
Record Dates: First submitted 2025-12-09; First posted 2025-12-12 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: HIV (Human Immunodeficiency Virus)
Keywords: HIV; emergency room; implementation science; machine-learning algorithm
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Emergencies | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Predictive Emergency Room Alerts (perA)Implementation Strategy (Active Comparator): Refers to patients within Care Management Agencies that have been randomized to use the pERA implementation strategy to delivery CCM/CC during that study period.
  Interventions: Other: predictive emergency room alerts (pERA)
- Standard of Care Implementation Strategy (Other): Refers to patients in Care Management Agencies that have been randomized to use their standard of care implementation strategy to deliver CCM/CC during that study period.
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: predictive emergency room alerts (pERA) — pERA is a machine-learning algorithm-driven implementation strategy that identifies patients at higher risk of emergency room visits and alerts the care manager to follow-up with them.
  Arms: Predictive Emergency Room Alerts (perA)Implementation Strategy
Other: Standard of care — Care managers interact with patients according to their standard of care protocols
  Arms: Standard of Care Implementation Strategy

SUMMARY:
This study tests a strategy for helping Care Management Agencies prioritize patients with HIV (PWH) for outreach and support. Under the new strategy, care managers are given a list of highest-priority patients who have been identified by a computer algorithm as being at high risk of going to the emergency room in the next two weeks. This strategy is compared to traditional (standard of care) care management, in which care managers reach out to patients based on a set schedule and their clinical judgement (but not based on a computerized report). We are looking at whether the use of the computer report helps care managers reach the right patients at the right time, preventing them from having to go to the emergency room.

DETAILED DESCRIPTION:
Comprehensive Care Management and Care Coordination (CCM/CC) is a medical case management intervention with demonstrated effectiveness in reducing ED visits and hospitalization for PWH, and improving both health outcomes (viral load, CD4 count) and retention in care. However, despite CCM/CC's effectiveness, there are persistent challenges to its implementation. This project is based on the scientific premise that the effectiveness of the CCM/CC intervention can be greatly improved by utilizing a data-driven implementation strategy that optimizes timely provision of CCM/CC services to the patients who need it most. Our community-based collaborator, Comprehensive Care Management Partners (CCMP) Health Home, has developed and validated a machine-learning algorithm that can reliably predict which of its PWH patients are most likely to visit the ED in the next two weeks. In this project, we will apply this algorithm as a targeted implementation strategy for CCM/CC, focusing service provision on the PWH who need it most, when they need it most. Our core hypothesis (supported by preliminary studies data) is that this "just-in-time" strategy for implementing a care management intervention will overcome both provider-level barriers to the provision of CCM/CC services and patient-level barriers to the receipt of HIV treatment and care. We will conduct a Hybrid 2 implementation-effectiveness trial, guided by the RE-AIM implementation science framework and the behavioral economics theory of Scarcity to collect rigorous data on the impact of this algorithm-driven implementation strategy on the reach, effectiveness, adoption, implementation and maintenance of the CCM/CC intervention

ELIGIBILITY:
Inclusion Criteria:

* Participants must be members of one of the Care Management Agencies that comprise the Community Care Management Partners (CCMP) Health Home
* Participants must be living with HIV

Exclusion Criteria:

* None, other than those listed above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2600 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
ER visits | Each 18 month cluster period (36 months total)
  Number of ER visits made by patients
Hospitalizations | Each 18 month Cluster Period (36 months total)
  Number of days of Hospitalization
Viral Suppression | Each 18 month cluster period (36 months total)
  Number of timepoints at which patient was virally suppressed
CD4 Count | Each 18 month Cluster Period (36 months total)
  CD4 Level at each data collection timepoint

CONTACTS AND LOCATIONS:
Overall Officials: Sarit A. Golub, PhD, MPH, Principal Investigator — Hunter College of The City University of New York
Locations (1):
- Community Care Management Partners Health Home, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
State health department requirements regarding these electronic medical record data prohibit sharing IPD.